CLINICAL TRIAL: NCT04410185
Title: Pain of Patients, Suffering of Caregivers: Evaluation of the Benefit of Full Consciousness Meditation in Oncology to Improve Stress and Quality of Life With Joint Participation of "Witness / Patient / Caregivers"
Brief Title: Pain of Patients, Suffering of Caregivers: Evaluation of the Benefit of Full Consciousness Meditation in Oncology
Acronym: IMPLIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Francois Baclesse (Other)
Collaborators: Fondation de France (Other); Cancéropôle Nord-Ouest (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2020-A00485-34
Record Dates: First submitted 2020-05-27; First posted 2020-06-01 (Actual); Last update posted 2021-03-04 (Actual); Status verified 2021-03

CONDITIONS: Cancer; Pain
Keywords: meditation; caregivers; patients with cancer
MeSH Terms: conditions — Neoplasms; Pain | interventions — Meditation

STUDY DESIGN:
Intervention Model Description: 3 separate populations will be recruited: Patients (n=10), caregivers (n=10), and control subjects (n=10)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MEDITATION (Experimental): Meditation sessions will take place over 12 weekly sessions of 1.5 hours. A retreat (3 hours) will be realized after the 9th session
  Interventions: Behavioral: Meditation

INTERVENTIONS:
Behavioral: Meditation — Meditation sessions will take place over 12 weekly sessions of 1.5 hours

SUMMARY:
The study is based on the realization of a meditation program associating patients, caregivers and control subjects

ELIGIBILITY:
Inclusion criteria for all participants (patients, caregivers and control subjects)

* Participants aged 18 or over
* Curious and motivated participant to participate in the program
* Participant with no current or previous experience of regular or intensive practice of meditation or a comparable practice. The practice is considered regular and / or intensive if:

  * it occurs more than one day per week for more than 6 consecutive months over the last 10 years,
  * and / or in case of more than 5 consecutive days of intensive practice (internship or retirement) in the last 10 years,
  * and / or more than 25 consecutive days of (cumulative) retirement over the last 10 years.
* Participant available to follow the full meditation program (3 month period)
* Participant agreeing to participate by signing the study information note
* Participant able to understand, speak and read French
* Patient capable of using digital media and having an internet connection

Patient-specific criteria (target population)

* Patients with cancer,
* State of health compatible with the study meditation program
* Patient affiliated to a social Health sytem

Caregiver-specific criteria

* All medical and / or paramedical staff of the sponsor Center in contact with patients (doctors, nurse, caregiver, radiotherapy manipulator MERM)

Criteria specific to the control population - Any voluntary person not belonging to the two categories above

Exclusion Criteria:

For all participants

* Participant with significant vulnerability factors dependence on alcohol and drugs, severe depression, severe social anxiety, recent mourning etc.).
* Participant who cannot submit to the follow-up of the trial for geographic, social or psychopathological reasons

For patients

* Very advanced stage of cancer disease with life-threatening commitment,
* Participant deprived of liberty or under guardianship

For control subjects

- Nursing staff, regardless of their place of practice

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2020-09-10 (Actual); Primary Completion 2021-02-11 (Actual); Study Completion 2021-02-11 (Actual)

PRIMARY OUTCOMES:
Evaluate the adherence of all participants to the full meditation program | 3 months after the beginning of program
  Proportion of participants adhering to the full meditation program (13 sessions)

CONTACTS AND LOCATIONS:
Locations (1):
- Centre François Baclesse, Caen, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Prevost V, Tran T, Clarisse B, Leconte A, Duchange N, Moutel G, Gouriot M. Shared Meditation Involving Cancer Patients, Health Professionals and Third Persons: Perceptions of Participants Through a Focus Group Study. Integr Cancer Ther. 2023 Jan-Dec;22:15347354231186995. doi: 10.1177/15347354231186995. PMID 37452577
- [Derived] Prevost V, Lefevre-Arbogast S, Leconte A, Delorme C, Benoit S, Tran T, Clarisse B. Shared meditation involving cancer patients, health professionals and third persons is relevant and improves well-being: IMPLIC pilot study. BMC Complement Med Ther. 2022 May 18;22(1):138. doi: 10.1186/s12906-022-03599-w. PMID 35585593
- [Derived] Prevost V, Clarisse B, Leconte A, Delorme C, Benoit S, Tran T. Meditation involving people with cancer, medical staff and witnesses: a pilot study exploring improvement in wellness and connectedness. BMJ Open. 2021 Nov 12;11(11):e048164. doi: 10.1136/bmjopen-2020-048164. PMID 34772746